CLINICAL TRIAL: NCT03904550
Title: Reversal of Neuromuscular Blockade in Patients With Severe Renal Impairment
Brief Title: Neuromuscular Blockade in Patients With Severe Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2018-0411
Record Dates: First submitted 2019-02-21; First posted 2019-04-05 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Neuromuscular Blockade; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — cisatracurium; Neostigmine; Rocuronium; Sugammadex

STUDY DESIGN:
Intervention Model Description: single site, randomized, controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cisatracurium + Neostigmine (Active Comparator): Patients in the cisatracurium/neostigmine group will receive 0.2 mg/kg of cisatracurium for neuromuscular paralysis during induction. Additional cisatracurium will be given to keep the patient at a neuromuscular depth of 1 twitch throughout the surgery until the last 30 minutes, during which the patient will be kept at 2 twitches.
  Interventions: Drug: Cisatracurium + Neostigmine
- Rocuronium + Sugammadex (Active Comparator): Patients in the rocuronium/sugammadex group will receive 0.6 mg/kg of rocuronium for neuromuscular paralysis during induction. Additional rocuronium will be given to keep the patient at a neuromuscular depth of 1 twitch throughout the surgery until the last 30 minutes, during which the patient will be kept at 2 twitches.
  Interventions: Drug: Rocuronium + Sugammadex

INTERVENTIONS:
Drug: Cisatracurium + Neostigmine — Maintenance neuromuscular blockade with boluses of cisatracurium to keep train-of-four (TOF) 1-2 twitches. For reversal, neostigmine with glycopyrrolate
  Arms: Cisatracurium + Neostigmine
Drug: Rocuronium + Sugammadex — Maintenance neuromuscular blockade with boluses of rocuronium to keep TOF 1-2 twitches. For reversal, sugammadex
  Arms: Rocuronium + Sugammadex

SUMMARY:
This study is intended to be a single-site, prospective, randomized, double-blinded study that intends to enroll a total of 60 patients with severe renal impairment undergoing surgery with general endotracheal anesthesia at Parkland Hospital. Patients will be randomized to receive either neostigmine (for reversal of cisatracurium) or sugammadex (for reversal of rocuronium). A standardized anesthetic protocol that is usual and customary for the type of operation the patient is having will be provided to the anesthesia teams of enrolled subjects. The remainder of the anesthetic care of the subject will not deviate from the standard of care. All patients will be monitored with continuous pulse oximetry postoperatively for 24 hours.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double-blinded study of surgical patients with severe renal impairment that seeks to address the following:

Specific Aim:

To determine whether rocuronium-induced moderate neuromuscular blockade and reversal with sugammadex achieves recovery of neuromuscular function (TOF ≥ 0.9) faster than reversal of cisatracurium-induced moderate neuromuscular blockade and reversal with neostigmine in patients with severe renal impairment.

Primary Hypothesis:

Patients with severe renal impairment who are reversed with sugammadex after rocuronium will achieve a TOF ≥0.9 within a time frame that is one-third of the time it takes for reversal with neostigmine after cisatracurium.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Severe renal impairment (CrCl < 30 mL/min)
* Undergoing non-emergent surgery that requires neuromuscular blockade
* Planned extubation in the operating room immediately after surgery
* American Society of Anesthesiologists (ASA) physical status classification 3 to 4
* Willing and able to consent in English or Spanish
* No personal history of neuromuscular disease

Exclusion Criteria:

* Age less than 18 or older than 80
* Patient does not speak English or Spanish
* Planned postoperative intubation/ventilation
* Allergy to sugammadex, neostigmine, glycopyrrolate, cisatracurium, or rocuronium
* Family or personal history of malignant hyperthermia
* Patient refusal
* Pregnant or nursing women
* "Stat" (emergent) cases
* Pre-existing muscle weakness of any etiology
* Patients on toremifene (a selective estrogen receptor modulator)
* Women on oral contraceptives who do not wish to use a non-hormonal method of contraception for 7 days following surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisatracurium + Neostigmine | Rocuronium + Sugammadex
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisatracurium + Neostigmine | Rocuronium + Sugammadex | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 14 | 22 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 11 | 21
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Time Until Complete Reversal of Neuromuscular Blockade
Description: Measure how long it takes to return from a TOF of 2 to a TOF ≥ 0.9.
Time Frame: In the operating room, the amount of time after administration of the reversal syringe to reach recovery of neuromuscular function (TOFR ≥ 90%) assessed up to 30 minutes.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cisatracurium + Neostigmine | Rocuronium + Sugammadex
Number analyzed (Participants) | 23 | 26
Minutes | 14.8 (6.1) | 3.5 (1.6)

ADVERSE EVENTS:
Time Frame: Up to post operative day 30
Arm/Group | Cisatracurium + Neostigmine | Rocuronium + Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03904550/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT03904550/ICF_001.pdf